CLINICAL TRIAL: NCT01790360
Title: Seek, Test, and Retain. Linkages for Black HIV+, Substance-Using Men Who Have Sex With Men.
Brief Title: Seek, Test, and Retain. Linkages for Black HIV+, Substance-Using MSM
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAI1585; 1R01DA032100-01 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-02-13 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Substance Abuse; Sexual Behavior
Keywords: MSM; HIV; Substance Abuse; Sexual Behavior
MeSH Terms: conditions — Substance-Related Disorders; Sexual Behavior | interventions — Patient Navigation; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigation (PN) (Active Comparator): Behavioral Intervention: 'Patient Navigation (PN) Intervention' participants will receive support from navigators in choosing a provider and remembering to attend appointments
  Interventions: Behavioral: Patient Navigation (PN) Intervention
- Financial Incentives (FI) (Experimental): Behavioral Intervention: 'Financial Incentives (FI) Intervention' participants will receive gift cards and money for attending clinic visits
  Interventions: Behavioral: Financial Incentives (FI) Intervention

INTERVENTIONS:
Behavioral: Patient Navigation (PN) Intervention — Patient Navigation is defined as an individual relationship between a navigator and participant to promote retention in the continuum of HIV care . For this study, three experienced navigators will be hired. Their primary role will be to ensure that participants are linked to an HIV primary care provider, that they attend at least one scheduled visit within three months of receiving a confirmed HIV diagnosis, and that they are retained in care (as defined by attending three HIV visits within nine months of diagnosis). To promote linkage to HIV care, navigators will help participants identify material and other barriers to accessing care and will work with participants to overcome those barriers.
  Other Names: PN Intervention; PN
  Arms: Patient Navigation (PN)
Behavioral: Financial Incentives (FI) Intervention — After confirmation that they have completed their first HIV primary care visit, Financial Incentive participants will receive a gift card. Additionally, the coordinator will flip a coin and give participants a bonus gift card if the coin flip comes up heads. Participants who attend the second HIV primary care visit will receive a gift card. Patients who attend a third HIV primary care visit will receive a gift card. Study staff will be responsible for confirming participants' attendance at appointments.
  Other Names: FI Intervention; FI
  Arms: Financial Incentives (FI)

SUMMARY:
The study will seek and recruit substance-using Black Men who have Sex with Men (MSM) in New York City for Human Immunodeficiency Virus (HIV) testing and will link and retain those who are HIV infected in HIV primary care. The STAR study has two primary objectives: to evaluate the feasibility and effectiveness of Respondent Driven Sampling (RDS) in the substance using Black MSM population for identifying individuals who are HIV infected and not in care; and to assess the relative effectiveness of patient navigation and financial incentives in linkage and retention to HIV care.

DETAILED DESCRIPTION:
The HIV epidemic in the United States most severely affects men who have sex with men (MSM): 61% of all new infections occur in this population. Black MSM bear a disproportionate burden, with prevalence of 28%, in contrast to 19% in MSM overall. Black MSM undergo HIV testing less frequently than other MSM; are less likely to be aware that they are HIV infected; are more likely to experience delays in entry into HIV care; and are less likely to be prescribed antiretroviral therapy (ART) when eligible. These disparities are pronounced in substance-using MSM, as substance users are at elevated risk of late diagnosis and delayed engagement in HIV care. The combination of pervasive stigma associated with MSM behavior and high rates of substance use hinders effective prevention efforts in this population, even as the prevalence of infection in Black MSM in some US cities approaches 50%. Reducing HIV-related disparities in MSM and among Black Americans are National HIV/AIDS Strategy priorities and are essential to the effort to control and prevent HIV/AIDS in the US.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black, African American, Caribbean Black, or multi-ethnic Black
* Identify as male
* Greater than 18 years old
* Have had sex with a man during the preceding 12 months
* Have ever used illicit drugs or alcohol to intoxication

Exclusion Criteria:

*Participation in other study assessing linkage and retention in HIV care

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1930 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Retention Rate (Linkage to Care) | Up to 3 months from HIV diagnosis
  Linkage to care will be defined as the attendance of at least one scheduled HIV primary care visit within three months of receiving a confirmed HIV diagnosis. Retention in care will be defined as three visits within nine months of HIV diagnosis.

SECONDARY OUTCOMES:
Dollars per patient linked and retained in care | Up to 9 months
  We will calculate dollars per patient linked and retained in care to measure cost-effectiveness of the two linkage/retention interventions: costs administering the incentives for the financial incentives arm and staffing costs for the peer navigation arm. All such values will then be adjusted by the opportunity cost of each participant's time. In addition, we will include fixed costs (eg, pamphlets and teaching materials to train the navigators) and the cost of space required to host the navigators.
Proportion of substance-using Black MSM who are recruited | Up to 3 years
  Effectiveness of Respondent-Driven Sampling (RDS) for seeking and recruiting substance-using Black MSM: the characteristics of RDS will be estimated using conventional proportion calculations, with confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa M El-Sadr, MD, Principal Investigator — Columbia University
Locations (1):
- Harlem Prevention Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Franks J, Mannheimer SB, Hirsch-Moverman Y, Hayes-Larson E, Colson PW, Ortega H, El-Sadr WM. Multiple strategies to identify HIV-positive black men who have sex with men and transgender women in New York City: a cross-sectional analysis of recruitment results. J Int AIDS Soc. 2018 Mar;21(3):e25091. doi: 10.1002/jia2.25091. PMID 29537178